CLINICAL TRIAL: NCT00047970
Title: The Sister Study: Genetic and Environmental Risk Factors for Breast Cancer
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Dale Sandler, Chief, Epidemiology Branch, DIR, National Institute of Environmental Health Sciences (NIEHS)
Other Study IDs: 02-E-N-271; NCT00339820 (obsolete NCT alias)
Record Dates: First submitted 2002-10-23; First posted 2002-10-24 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2012-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Sisters
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Sister Study is prospectively examining environmental and familial risk factors for breast cancer and other diseases in a cohort of 50,884 sisters of women who have had breast cancer. Such sisters have about twice the risk of developing breast cancer as other women.

DETAILED DESCRIPTION:
The Sister Study is prospectively examining environmental and familial risk factors for breast cancer and other diseases in a cohort of 50,884 sisters of women who have had breast cancer. Such sisters have about twice the risk of developing breast cancer as other women. The frequency of any relevant genes and shared risk factors will also be higher. Studying sisters enhances our ability to understand the interplay of genes and environment in breast cancer risk and to identify potentially preventable risk factors. We assess exposures before the onset of disease, thus avoiding biases common to retrospective studies. The assembled cohort has created a framework from which to test new hypotheses as they emerge.

Cancer-free sisters aged 35-74 were recruited nationally. Enrollment was completed July 2009 with 50,884 women fully enrolled. Participants have enrolled from all 50 states and Puerto Rico. The cohort is now being followed actively. Cohort members are occasionally invited to participate in add-on studies, which sometimes include asking participants to invite their family members to provide information.

Data on potential risk factors and current health status were collected with telephone interviews and self-completed questionnaires. Blood, urine, and environmental samples were collected and banked for future use in nested studies of women who develop breast cancer (or other diseases) and a sample of those who don't. The cohort is being followed prospectively for 10 or more years. Annual questionnaires update medical history and changes in exposures. About 300 new cases of breast cancer are expected to occur in the cohort each year. Analyses are ongoing and assess the independent and combined effects of environmental exposures and genetic polymorphisms that affect estrogen metabolism, DNA repair, and response to specific environmental exposures. Future analyses will focus on known and potential risk factors (e.g. smoking, occupational exposures, alcohol, diet, obesity) and include measurement of phthalates, phytoestrogens, insulin, growth factors, micro-nutrients, and genes. Women who develop breast cancer during the study are followed to assess the role of environment and genes in healthy survival following diagnosis and treatment. The cohort will also be used to explore risk for other diseases (e.g. heart disease, osteoporosis, other hormonal cancers, and autoimmune diseases) that are important for women.

ELIGIBILITY:
Inclusion Criteria:

Women who are eligible for the Sister Study:

* Have a sister (living or deceased) who had breast cancer
* Ages 35-74
* Never had breast cancer themselves
* Live in the United States

The Sister Study is currently recruiting sisters of women diagnosed with breast cancer nationwide.

Ages: 35 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50884 (Actual)
Dates: Start 2003-08; Primary Completion 2009-08 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NIEHS, Research Triangle Park, North Carolina, United States

REFERENCES:
- [Derived] O'Brien KM, Sandler DP. Reply to "Vitamin D and breast cancer: Stop torturing the data!". Cancer. 2022 Aug 1;128(15):3000-3001. doi: 10.1002/cncr.34274. Epub 2022 Jun 1. No abstract available. PMID 35647759
- [Derived] Kresovich JK, Park YM, Keller JA, Sandler DP, Taylor JA. Healthy eating patterns and epigenetic measures of biological age. Am J Clin Nutr. 2022 Jan 11;115(1):171-179. doi: 10.1093/ajcn/nqab307. PMID 34637497
- [Derived] Petimar J, Park YM, Smith-Warner SA, Fung TT, Sandler DP. Dietary index scores and invasive breast cancer risk among women with a family history of breast cancer. Am J Clin Nutr. 2019 May 1;109(5):1393-1401. doi: 10.1093/ajcn/nqy392. PMID 30968114
- See also: Sister Study Website — http://www.sisterstudy.org